CLINICAL TRIAL: NCT06482112
Title: A Phase 2a Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Different Dosing Regimens of Efinopegdutide (MK-6024) in Adults With Metabolic Dysfunction-Associated Steatotic Liver Disease
Brief Title: Alternate Dosing Study of MK-6024 in Adults With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) (MK-6024-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6024-016; MK-6024-016 (Other: MSD)
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Non-alcoholic Fatty Liver Disease; Nonalcoholic Fatty Liver Disease; Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Efinopegdutide Q1W 10 mg (Active Comparator): Participants will receive efinopegdutide Q1W via subcutaneous (SC) injection for 28 weeks in a dose-escalating regimen of 2 mg for 4 weeks, 4 mg for 4 weeks, 7 mg for 4 weeks, and 10 mg for up to 16 weeks.
  Interventions: Drug: Efinopegdutide
- Efinopegdutide Q2W 10 mg (Experimental): Participants will receive efinopegdutide Q2W via SC injection for 28 weeks in a dose-escalating regimen of 2 mg for 4 weeks, 4 mg for 4 weeks, 7 mg for 4 weeks, and 10 mg for up to 16 weeks.
  Interventions: Drug: Efinopegdutide
- Efinopegdutide Q2W 15 mg (Experimental): Participants will receive efinopegdutide Q2W via SC injection for 28 weeks in a dose-escalating regimen of 2 mg for 4 weeks, 4 mg for 4 weeks, 7 mg for 4 weeks, 10 mg for 4 weeks, and 15 mg for up to 12 weeks.
  Interventions: Drug: Efinopegdutide

INTERVENTIONS:
Drug: Efinopegdutide — SC injections in dose-escalation regimens potentially including doses of 2 mg, 4 mg, 7 mg, and 10 mg in all arms and 15 mg in the Efinopegdutide Q2W 15 mg arm
  Other Names: MK-6024; HM12525A; JNJ-64565111

SUMMARY:
This study will evaluate the effect of efinopegdutide administration once every 2 weeks (Q2W) versus once weekly (Q1W) on mean relative reduction from baseline in liver fat content (LFC) after 28 weeks, as well as the safety and tolerability of the different regimens of efinopegdutide.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has body mass index (BMI) ≥25 kg/m^2 (≥23 kg/m^2 for Asian participants) AND has stable weight, defined as ≤5% gain or loss of body weight for at least 3 months before screening
* Has no history of type 2 diabetes mellitus (T2DM) OR has a history of T2DM with a glycated hemoglobin (A1C) ≤9% AND the T2DM is controlled by diet or stable doses of oral antihyperglycemic agents (AHAs)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following

* Has a history or evidence of chronic liver disease other than Metabolic dysfunction-associated steatotic liver disease (MASLD) or Metabolic dysfunction-associated steatohepatitis (MASH)
* Has evidence of decompensated liver disease including, but not limited to ascites, esophageal or gastric variceal bleeding, hepatocellular carcinoma, hepatic encephalopathy, splenomegaly, or spontaneous bacterial peritonitis
* Has a history of pancreatitis
* Has a history of type 1 diabetes mellitus (T1DM), diabetic ketoacidosis, or diabetes secondary to pancreatectomy.
* Has symptomatic hyperglycemia
* Has a history of a bariatric surgical procedure ≤5 years before Screening or a known clinically significant gastric emptying abnormality
* Has a history of obesity with a known secondary cause
* Has significant systemic or major illnesses, including recent (≤6 months before Screening) onset of events of congestive heart failure, unstable angina, myocardial infarction, arterial revascularization, stroke, or transient ischemic attack
* Is unable to have Magnetic Resonance Imaging-Estimated Proton Density Fat Fraction (MRI-PDFF) due to: Claustrophobia to a degree that prevents tolerance of an MRI-PDFF scanning procedure. Note: Sedation is permitted, at the discretion of the investigator; Metallic implants that prevent MRI-PDFF examination; Exceeds the body habitus and/or weight limitations for the MRI scanner

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Mean relative reduction from baseline in liver fat content (LFC) at Week 28 | Baseline and Week 28
  LFC will be measured with liver images taken by Magnetic Resonance Imaging Estimated Proton Density Fat Fraction (MRI-PDFF) and analyzed by blinded independent central review (BICR). Relative Reduction from Baseline to Week 28 = (Baseline - Week 28) / Baseline x 100%. Mean relative reduction from baseline in LFC will be presented.
Percentage of participants who experienced an adverse event (AE) | Up to Week 32
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants who experienced an AE will be presented.
Percentage of pariticpants who discontinued study intervention due to an AE | Up to Week 28
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants who discontinued study intervention due to an AE will be presented.

SECONDARY OUTCOMES:
Mean percent change from baseline in body weight at Week 28 | Baseline and Week 28
  Body weight in kilograms will be measured using a standardized, digital scale. The mean percent change from baseline in body weight after 28 weeks will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp and Dohme LLC
Locations (39):
- United States (36):
  - The Institute for Liver Health II dba Arizona Clinical Trial-The Institute for Liver Health ( Site 0, Chandler, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health - Peoria ( Site 0224), Peoria, Arizona
  - Arizona Liver Health ( Site 0211), Tucson, Arizona
  - Del Sol Research Management, LLC ( Site 0209), Tucson, Arizona
  - Om Research LLC ( Site 0207), Camarillo, California
  - Gastroenterology and Liver Institute ( Site 0263), Escondido, California
  - Velocity Clinical Research, Gardena ( Site 0235), Gardena, California
  - Velocity Clinical Research, Huntington Park ( Site 0210), Huntington Park, California
  - California Liver Research Institute ( Site 0216), Pasadena, California
  - Acclaim Clinical Research ( Site 0241), San Diego, California
  - Velocity Clinical Research, Santa Ana ( Site 0250), Santa Ana, California
  - Velocity Clinical Research, Panorama City ( Site 0228), Van Nuys, California
  - Excel Medical Clinical Trials ( Site 0268), Boca Raton, Florida
  - AGA Clinical Trials ( Site 0274), Hialeah, Florida
  - Neoclinical Research ( Site 0275), Hialeah, Florida
  - Homestead Associates in Research, Inc. ( Site 0243), Homestead, Florida
  - Floridian Clinical Research, LLC ( Site 0208), Miami Lakes, Florida
  - Southeast Clinical Research Center ( Site 0223), Dalton, Georgia
  - Velocity Clinical Research Rockville ( Site 0245), Rockville, Maryland
  - The Machuca Foundation ( Site 0218), Las Vegas, Nevada
  - Excel Clinical Research, LLC ( Site 0200), Las Vegas, Nevada
  - Basil Clinical ( Site 0246), Inwood, New York
  - Lucas Research, Inc ( Site 0204), Morehead City, North Carolina
  - Texas Clinical Research Institute ( Site 0230), Arlington, Texas
  - Pinnacle Clinical Research ( Site 0203), Austin, Texas
  - Velocity Clinical Research, Austin ( Site 0201), Austin, Texas
  - Pinnacle Clinical Research-Corpus Christi ( Site 0267), Corpus Christi, Texas
  - Zenos Clinical Research ( Site 0240), Dallas, Texas
  - South Texas Research Institute ( Site 0226), Edinburg, Texas
  - Houston Research Institute ( Site 0221), Houston, Texas
  - American Research Corporation ( Site 0234), San Antonio, Texas
  - Clinical Trials of Texas, LLC-Clinical Research ( Site 0252), San Antonio, Texas
  - Pinnacle Clinical Research-Clinical Research Coordination ( Site 0229), San Antonio, Texas
  - Impact Research Institute ( Site 0227), Waco, Texas
  - Olympus Family Medicine/CCT Research ( Site 0266), Holladay, Utah
  - South Ogden Family Medicine/ CCT Research ( Site 0255), South Ogden, Utah
- Puerto Rico (3):
  - San Juan Bautista School of Medicine - Clinical Research Unit ( Site 0104), Caguas
  - Klinical Investigations Group-Clinical Research ( Site 0100), San Juan
  - Pan American Center for Oncology Trials - Ciudadela ( Site 0101), San Juan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com